CLINICAL TRIAL: NCT00244400
Title: Examine the Possible Association of Hepatic CYP3A Activity and the Susceptibility to Femur Head Necrosis
Status: Completed | Type: Observational
Sponsor: Osaka City University (Other)
Other Study IDs: 338
Record Dates: First submitted 2005-10-25; First posted 2005-10-26 (Estimated); Last update posted 2006-10-17 (Estimated); Status verified 2006-10

CONDITIONS: Femur Head Necrosis
Keywords: Femur Head Necrosis; CYP3A
MeSH Terms: conditions — Femur Head Necrosis

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The purpose of the present study was to examine the possible association of hepatic CYP3A activity and the susceptibility to femur head necrosis in patients treated with corticosteroids.

DETAILED DESCRIPTION:
Femur head necrosis is one of the major side effects of corticosteroid therapy. Since corticosteroids are metabolized by hepatic cytochrome P-450 (CYP) 3A, a low endogenous activity of this enzyme may contribute to the pathogenesis of ONFH. The purpose of the present study was to examine the possible association of hepatic CYP3A activity and the susceptibility to femur head necrosis in patients treated with corticosteroids.

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis of avascular necrosis of the femur

Exclusion Criteria:

* Old age (> 70 years)
* Severe hepatic or renal dysfunction
* Heart disease
* Current use of known CYP3A-inducing or -inhibiting drugs
* Morbid obesity

Ages: 14 Years to 70 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 200
Dates: Start 2002-11; Study Completion 2006-01

CONTACTS AND LOCATIONS:
Overall Officials: Yasunori Kaneshiro, M.D., Principal Investigator — Department of Orthopedic Surgery, Graduate School of Medicine, Osaka City University
Locations (1):
- Graduate School of Medicine, Osaka City University, Osaka, Osaka, Japan